CLINICAL TRIAL: NCT00298103
Title: Antibiotic Resistant Community-Acquired E. Coli
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: IRB# 0602065
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: E Coli Infection
Keywords: Antibiotic resistant; Infection
MeSH Terms: conditions — Escherichia coli Infections; Infections

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to review patients with E. coli infections at UPMC from January 1, 2004 to December 31, 2005 to determine if these infections have arisen in the community rather than in hospitals or nursing homes. The occurrence of such resistant isolates could be devastating if they were associated with bloodstream infection, such as sometimes accompanies urinary tract infection, since antibiotic resistant E. coli is not suspected in isolates coming from the community.

DETAILED DESCRIPTION:
The following variables will be followed: age, sex, hospital location at the time of positive culture (ER, medical ward, ICU etc), prior hospitalization or nursing home admission, receipt of outpatient dialysis or other regular medical care (eg, outpatient chemotherapy), presence of invasive devices, receipt of antibiotics, including their type and whether they were adequate for the resistance profile of the organism, prior positive microbiologic cultures.

ELIGIBILITY:
Inclusion Criteria:

* ll patients with E. coli infections during the time period of the study will be reviewed. A community-associated E. coli isolate will be defined as one which was recovered from a clinical culture from a patient at UPMC-P who had no established risk factors for infection with an antibiotic resistant organism.

Established risk factors are defined as:

* Isolation of the organism two or more days after admission for hospitalization OR A history of hospitalization, surgery, dialysis, or residence in a long-term care facility within one year before the culture date
* OR The presence of an indwelling catheter or percutaneous medical device (eg, tracheostomy tube, gastrostomy tube, or Foley catheter) at the time of the culture
* OR Previous isolation of an antibiotic resistant organism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with e coli infections
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States